CLINICAL TRIAL: NCT04987515
Title: Clinical Evaluation of Fenestration Decompression Combined With Secondary Curettage for Ameloblastoma of the Jaw: Retrospective Radiographic Analysis
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, hejie, associate chief physician, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: 123456
Record Dates: First submitted 2021-07-30; First posted 2021-08-03 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Cystic Cavity Area Reduction Efficiency; the Recurrence of the Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fenestration decompression combined with secondary curettage (FDSC): Design of the opening window reasonably；Making cyst plug；secondary curettage
  Interventions: Procedure: fenestration decompression combined with secondary curettage
- local curettage (LC): The tumor was removed by local curettage only

INTERVENTIONS:
Procedure: fenestration decompression combined with secondary curettage — First，fenestration decompression was performed. then, patients return every 3 months for follow up. If the cystic cavity area was gradually reduced after one year of follow-up, patients should be considered for secondary curettage surgery.
  Groups: Fenestration decompression combined with secondary curettage (FDSC)

SUMMARY:
Objectives: To investigate the outcomes of fenestration decompression combined with secondary curettage (FDSC) in the surgical treatment of jaw ameloblastoma.

Methods: Medical records of patients diagnosed as multicystic ameloblastoma (MA) or unicystic ameloblastoma (UA) by routine pathology were collected from January 2010 to December 2017 in Ninth People's Hospital, Shanghai JiaoTong University Medical College. Patients were divided into two groups based on the management regimen: FDSC group, and local curettage (LC) group. Patients were followed up for 3-8 years, using panoramic radiography to measure the change of the area of the cystic cavity involved in ameloblastoma and the recurrence or malignant transformation of the tumor in both groups. A total of 233 eligible patients were selected for provisional screening, including 145 patients with MA, and 88 patients with UA.

ELIGIBILITY:
Inclusion Criteria:

-Medical records of patients who were diagnosed with multicystic ameloblastoma (MA) or unicystic ameloblastoma (UA) by routine pathology were collected from January 2010 to December 2017 in Ninth People's Hospital of Shanghai JiaoTong University Medical College.

Exclusion Criteria:

* followed up less than 3 years
* For FDSC group, fenestration decompression failed
* recurrent ameloblastoma
* received other type of surgery;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical records of patients diagnosed as multicystic ameloblastoma (MA) or unicystic ameloblastoma (UA) by routine pathology were collected from January 2010 to December 2017 in Ninth People's Hospital, Shanghai JiaoTong University Medical College. Patients were divided into two groups based on the management regimen: fenestration decompression combined with secondary curettage (FDSC) group, and local curettage (LC) group. Patients were followed up for 3-8 years, using panoramic radiography to measure the change of the area of the cystic cavity involved in ameloblastoma and the recurrence or malignant transformation of the tumor in both groups.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Cystic cavity area reduction efficiency | 3 years after surgery
  (good effect case number + moderate effect case number)/total case number

SECONDARY OUTCOMES:
Tumor recurrence rate | 3 years after surgery
  the recurrence case number/total case number

OTHER OUTCOMES:
malignant transformation rate | 3 years after surgery
  malignant transformation case number/total case number

IPD SHARING:
Plan to Share IPD: Undecided